CLINICAL TRIAL: NCT02766283
Title: Observational Study on Hypothyroidism in Young Children Following Iodine Contrast Exposure
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18614
Record Dates: First submitted 2016-05-06; First posted 2016-05-09 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Hypothyroidism
Keywords: Children; Iodinated contrast agents
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Iodinated contrast agents: children age 0-3 years (inclusive), who underwent a iodine contrast enhanced radiological examination.
  Interventions: Drug: iodinated contrast agents

INTERVENTIONS:
Drug: iodinated contrast agents — Intravascular application

SUMMARY:
To investigate the incidence of detected hypothyroidism after iodinated contrast exposure in pediatric patients from birth to 3 years of age (inclusive) in a routine clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

- All children age 0-3 years (inclusive) who are identified of having undergone a radiological examination with intravascular use of an iodinated contrast agent.(e.g.

contrast enhanced CT, cardioangiography)

Exclusion Criteria:

* Congenital Hypothyroidism or other forms of preexisting hypothyroidism
* Preexisting thyroid hormone replacement therapy less than three months of observation before the radiological examination (if greater than three months old)
* Less than two weeks follow-up available after the contrast exposure.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Members of Maccabi Health Services database (Israel)
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a retrospective cohort study, using the data from the years 1998 until 2015 in the database of Maccabi Health Services (Israel).
Pre-assignment Details: Between 1.1.1998 and 31.12.2015, 877 participants were identified. After applying exclusion criteria, 34 participants were excluded from the initial cohort and the final cohort consisted of 843 participants.
Groups:
- Iodine Contrast Agent: The data used for this retrospective cohort study was from the years 1998 until 2015. The study population consisted of children ages 0-3 (inclusive) who have undergone a radiological examination with an iodinated contrast agent (contrast enhanced CT and cardio-angiography). Follow-up for the outcome (hypothyroidism) was for up to one year after contrast exposure. Incident cases of hypothyroidism were detected by: thyroid-stimulating hormone (TSH) levels, coded diagnosis of hypothyroidism or start of new thyroid replacement therapy.
Period: Overall Study
Arm/Group | Iodine Contrast Agent
Started | 843
Completed | 816
Not Completed | 27
Not completed — Lost to Follow-up | 27

BASELINE CHARACTERISTICS:
Population: Final Cohort
Groups:
- Iodine Contrast Agent: The data used for this retrospective cohort study was from the years 1998 until 2015. The study population consisted of children ages 0-3 (inclusive) who have undergone a radiological examination with an iodinated contrast agent (contrast enhanced CT and cardio-angiography). Follow-up for the outcome (hypothyroidism) was for up to one year after contrast exposure. Incident cases of hypothyroidism were detected by: TSH levels, coded diagnosis of hypothyroidism or start of new thyroid replacement therapy.
Arm/Group | Iodine Contrast Agent
Number analyzed (Participants) | 843
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.06 (0.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 382
  Male | 461
Weight [Mean (Standard Deviation); unit: Kilograms] | 8.80 (3.39)
Comorbidity [Number; unit: Participants]
  Cardio | 495
  Diabetes | 1
  Cancer | 21
  Overweight | 12
Sum of Examinations [Count of Participants; unit: Participants]
  1 | 775
  >= 2 | 68
Type of 1st examination [Count of Participants; unit: Participants]
  Cardio-angiography | 481
  CT | 362
Type of >=2nd examination [Count of Participants; unit: Participants] — Population: Participants in final cohort who underwent the 2nd examination
  Participants
    number analyzed (Participants) | 68
    Cardio-angiography | 47
    CT | 21
Time between examinations [Mean (Standard Deviation); unit: Days]
  First and second | 282.79 (252.34)
  Second and third | 208.19 (180.01)
  Third and fourth | 212.00 (196.28)
Dispenses of hypothyroidism inducing drugs [Number; unit: Participants]
  Anticonvulsants | 21
  Amiodarone | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Pediatric Patients With Detected Hypothyroidism After Iodinated Contrast Exposure in a Routine Clinical Practice Setting
Time Frame: Up to one year after iodinated contrast material (ICM) exposure (828 person years)
Population: Final Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Iodine Contrast Agent
Number analyzed (Participants) | 843
Participants | 11

2. Secondary Outcome: Baseline Characteristics (Sex) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Final Cohort
Measure: Count of Participants; unit: Participants
Groups:
- No Hypothyroidism Indication: Participants without potential hypothyroidism detected during the one-year follow up period (828 person years)
- Hypothyroidism Indication: Participants with potential hypothyroidism detected during the one-year follow up period (828 person years)
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Participants
  Male | 454 | 7
  Female | 378 | 4

3. Secondary Outcome: Baseline Characteristics (Age) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: At first examination
Population: Final Cohort
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Years | 1.07 (0.86) | 0.53 (0.96)

4. Secondary Outcome: Baseline Characteristics (Weight) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Within a range of ±360 days of the first examination
Population: Final Cohort
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Kilograms | 8.84 (3.37) | 6.57 (3.74)

5. Secondary Outcome: Baseline Characteristics (Comorbidity) of the Cases With Hypothyroidism and of the Rest of the Cohort
Time Frame: Prior to first examination
Population: Final Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Participants
  Cardio | 485 | 10
  Diabetes | 1 | 0
  Cancer | 21 | 0
  Overweight | 12 | 0

6. Secondary Outcome: Baseline Characteristics (Sum of Examinations) in Cases With an Indication of Hypothyroidism and Cases Without
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Final Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Participants
  1 | 765 | 10
  >=2 | 67 | 1
Statistical Analysis 1: Comparison: No Hypothyroidism Indication vs Hypothyroidism Indication; Test type: Superiority or Other; p = 0.90, Chi-squared

7. Secondary Outcome: Baseline Characteristics (Type of 1st Examination) in Cases With an Indication of Hypothyroidism and Cases Without
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Final Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Participants
  Cardio-angiography | 471 | 10
  CT | 361 | 1
Statistical Analysis 1: Comparison: No Hypothyroidism Indication vs Hypothyroidism Indication; Test type: Superiority or Other; p = 0.022, Chi-squared

8. Secondary Outcome: Baseline Characteristics (Type of 2nd Examination) in Cases With an Indication of Hypothyroidism and Cases Without
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Final Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Participants
  Cardio-angiography | 46 | 1
  CT | 21 | 0

9. Secondary Outcome: Baseline Characteristics (Time Between Examinations) in Cases With an Indication of Hypothyroidism and Cases Without
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Final Cohort
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | No Hypothyroidism Indication | Hypothyroidism Indication
Number analyzed (Participants) | 832 | 11
Days
  First and second: number analyzed (Participants) | 832 | 1
  First and second | 282.72 (254.24) | 288 (NA) — Only one participants underwent the second examination among the cases with an hypothyroidism indication
  Second and third: number analyzed (Participants) | 832 | 0
  Second and third | 208.19 (180.01) |
  Third and fourth: number analyzed (Participants) | 832 | 0
  Third and fourth | 212.00 (196.28) |

10. Secondary Outcome: Time-relation Between Iodine Contrast Exposure and Diagnosis of Hypothyroidism
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Final Cohort
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Final Cohort: Participants without potential hypothyroidism detected during the one-year follow up period (828 person years)
Arm/Group | Final Cohort
Number analyzed (Participants) | 828
Days | 76.54 (93.05)

11. Secondary Outcome: The Duration of Hypothyroidism Episode in the "Probable Iodine Induced" Category
Description: Based on the information collected from the database, the probable longest duration of Hypothyroidism was ascertained for the cases below.
Time Frame: Up to one year after ICM exposure (828 person years)
Population: Probable iodine-induced hypothyroidism: (N=8) included all potential cases of hypothyroidism with no other cause than the previous ICM exposure could be identified.
Measure: Number; unit: Months
Groups:
- Probable Iodine-induced Hypothyroidism: Included all potential cases of hypothyroidism with no other cause than the previous ICM exposure could be identified.
Arm/Group | Probable Iodine-induced Hypothyroidism
Number analyzed (Participants) | 8
Months
  Case number 2 | NA — Thyroid replacement therapy was dispensed
  Case number 3 | 2
  Case number 6 | NA — Thyroid replacement therapy was dispensed
  Case number 10 | 2

12. Secondary Outcome: The Duration of Hypothyroidism Episode in the "Probable Iodine Induced" Category
Description: Based on the information collected from the database, the probable shortest duration of Hypothyroidism was ascertained for the cases below.
Time Frame: Up to one year after ICM exposure (828 person years)
Population: as for outcome 11
Measure: Number; unit: Months
Arm/Group | Probable Iodine-induced Hypothyroidism
Number analyzed (Participants) | 8
Months
  Case number 4 | 4
  Case number 7 | 10

13. Secondary Outcome: The Duration of Hypothyroidism Episode in the "Probable Iodine Induced" Category
Description: as for outcome 12
Time Frame: Up to one year after ICM exposure (828 person years)
Population: as for outcome 11
Measure: Number; unit: Days
Arm/Group | Probable Iodine-induced Hypothyroidism
Number analyzed (Participants) | 8
Days
  Case number 5 | 14
  Case number 11 | 8

ADVERSE EVENTS:
Time Frame: Up to one year after contrast exposure.
Description: This study is a retrospective study using data from the database in Israel. The safety outcome focused on the incidence of hypothyroidism for up to one year after iodine contrast exposure, detected by: TSH levels, coded diagnosis of hypothyroidism or start of new thyroid replacement therapy. Please refer to the result of primary outcome measure.
Arm/Group | Iodine Contrast Agent
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study is a retrospective database analysis study. The safety outcome focused on the incidence of hypothyroidism for up to one year after iodine contrast exposure. Please refer to the result of primary outcome measure for safety evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other